CLINICAL TRIAL: NCT04738916
Title: The Impact of Low-intensity Whole-body Vibration Training on Extensor Muscles Strength, and Mechanical Properties of Lower Limb
Brief Title: Vibration Training in Healthy Individuals
Acronym: MusMechPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Filiz Basol, PT, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BEU
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Vibration; Exposure; Muscle Strength; Lower Limb
Keywords: muscle mechanical properties

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vibration Group (Experimental): The vibration group was included in the low frequency (25 Hz), low amplitude (2mm), fixed six-week training on two non-consecutive days of the week.
  Interventions: Device: Whole-body vibration training
- Control Group (No Intervention): No training was given to the control group.

INTERVENTIONS:
Device: Whole-body vibration training — Whole body vibration (WBV) is a form of treatment that has been shown to have an important role in increasing neuromuscular performance, improving muscular strength, balance. The technique involves standing and holding positions, or performing prescribed exercises, on a platform that is vibrating at a programmed frequency, amplitude, and magnitude of oscillationWhole-body vibration (WBV) is a therapeutic method that exposes the entire body to mechanical oscillations while the patient stands or sits on a vibrating platform.
  Arms: Vibration Group

SUMMARY:
The aim of the study was to examine the effect of six-week constant, low frequency and low amplitude Whole Body Vibration training on the strength and mechanical properties of the lower limb knee extensors and ankle joint dorsi flexor muscles.

DETAILED DESCRIPTION:
The aim of the study was to examine the effect of six-week constant, low frequency and low amplitude Whole Body Vibration training on the strength and mechanical properties of the lower limb knee extensors and ankle joint dorsi flexor muscles.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering
* Weight less than 120 kg

Exclusion Criteria:

* The presence of a history of trauma in the lower extremity in the last six months
* Limitation of movement in the lower extremity
* A history of cardiovascular, neurological, orthopedic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Muscle mechanical properties | at 6-week
  MyotonPRO evaluation: Non-invasive assessment of state of tension, biomechanical and viscoelastic properties of lower limb extensors.

SECONDARY OUTCOMES:
Muscle Strength | at 6-week
  Lafayette: Hand-held dynamometer evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University Sports Laboratory, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No